CLINICAL TRIAL: NCT01189006
Title: A Double-blind, Placebo-Controlled, Randomized Study of the Efficacy of Dextromethorphan as Add-On Therapy to Risperidone Versus Risperidone Alone in Patients With Schizophrenia
Brief Title: Add-On Therapy to Risperidonein Schizophrenia
Acronym: DM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM-Schizo; Taiwan NIH (Other Grant/Funding Number: DOH-95-TD-I-111-004)
Record Dates: First submitted 2010-08-23; First posted 2010-08-26 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2010-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dextromethorphan (Experimental): Research clinical trial of double-blind, stratified randomized, parallel group, double-centre study
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — Add-On double-blind study treatment commenced at randomization for 11 weeks while patients were continuing open-label risperidone. Randomization was immediately preceded by a one week open-label Risperidone-Only Treatment period. Patients who were receiving antipsychotics medication(s) at screen other than risperidone alone was withdrawn from previous non-risperidone medication(s) and at the same time commenced risperidone in titrating doses over a week. This Antipsychotic Switch-Over Period occurred between Screen and Risperidone-Only Treatment period. Patients remained hospitalized for at least during the Risperidone-Only treatment Period and first week of Add-On treatment Period.

SUMMARY:
These results suggest that the DA neuroprotection provided by DM in the inflammation-related neurodegenerative models is not mediated through the NMDA receptor.

DETAILED DESCRIPTION:
Liu et al. (2003) have reported that DM protected dopamine (DA) neurons against inflammation-mediated degeneration. Zhang et al.'s (2004) novel finding was that 1-10 μM DM protected DA neurons against LPS (10 ng/mL)-induced reduction of DA uptake functionally in rat primary mixed mesencephalic neuron-glia cultures. Morphologically, in lipopolysaccharide (LPS)-treated cultures, in addition to the reduction of abundance of DA neurons, the dendrites of the remaining DA neurons were significantly less elaborate than those of controls. In cultures pretreated with DM (10 μM) before LPS stimulation, DA neurons were significantly more numerous and the dendrites less affected. Significant neuroprotective was observed in cultures with DM added up to 60 minutes after the addition of LPS. Thus, DM significantly protects DA neurons not only with pretreatment but also with post-treatment (Zhang et al. 2004). The mechanism of the neuronprotective effect of DM is associated with the inhibition of microglia activation but not with its NMDA receptor antagonist property. Zhang et al. (2005) have examined several N-methyl-D-aspartate (NMDA) receptor antagonists, including MK801, AP5, and memantine. Results from these studies indicate that among these compounds tested there was no correlation between the affinity of NMDA receptor antagonist activity and potency of the neuroprotective on DA neurons. On the contrary, a better correlation was found between the anti-inflammatory potency and the neuron protection. These results suggest that the DA neuroprotection provided by DM in the inflammation-related neurodegenerative models is not mediated through the NMDA receptor. This conclusion is not in conflict with the previous reports, indicating that NMDA receptor blockade is associated with the neuroprotective effect of DM in acute glutamate-induced excitotoxicity models. The above evidences of benefit on auto-immune system with dextromethorphan would support that dextromethorphan as add-on therapy to atypical antipsychotics might be more effective than atypical antipsychotics alone on improvement of both positive and negative symptoms in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged ≧18 and ≦60 years.
2. A diagnosis of schizophrenia or schizoaffective disorder according to DSM-IV criteria made by a specialist in psychiatry.
3. Acute exacerbation of schizophrenia.
4. A total of PANSS score of at least 60 at screen.
5. History of schizophrenia ≦ 15 years (from onset of prodromal symptoms).
6. Signed informed consent by patient or legal representative
7. Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

1. Women of childbearing potential not using adequate contraception as per investigator judgement or not willing to comply with contraception for duration of study.
2. Less than a full cycle has lapsed at time of screening following the last injection of a depot antipsychotic
3. Females who are pregnant or nursing.
4. Patient has received dextromethorphan, or other selective cyclo- oxygenase 2 inhibitors, or other anti-inflammatory medication within 1 week prior to first dose of double-blind medication.
5. Axis-I DSM-IV diagnosis other than schizophrenia or schizoaffective disorder.
6. Current evidence of an uncontrolled and/or clinically significant medical condition, e.g., cardiac, hepatic and renal failure that in the judgement of the investigator, would compromise patient safety or preclude study participation.
7. History of intolerance to risperidone or dextromethorphan or other Cox-2 inhibitors.
8. History of sensitivity reaction (e.g., urticaria, angioedema, bronchospasm, severe rhinitis, anaphylactic shock) precipitated by dextromethorphan.
9. Patient has received electroconvulsive therapy (ECT) within 4 weeks prior to first dose of double-blind medication.
10. Diagnosis of or treatment for oesophageal, gastric, pyloric channel, or duodenal ulceration or related complications (bleeding and/or perforation) within 30 days prior to receiving first dose of double-blind medication.
11. Inclusion in another schizophrenia study or study for another indication with psychotropics within the last 30 days prior to start of study.
12. Increase in total SGOT, SGPT, gamma-GT, BUN and creatinine by more than 3X ULN (upper limit of normal).
13. History of idiopathic or drug-induced agranulocytosis.
14. Alcohol, illegal or other substance-abuse within 6 months prior to study start, as defined by DSM-IV criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
positive and negative symptoms in schizophrenia | baseline
positive and negative symptoms in schizophrenia | week1
positive and negative symptoms in schizophrenia | week2
positive and negative symptoms in schizophrenia | week4
positive and negative symptoms in schizophrenia | week6
positive and negative symptoms in schizophrenia | week8
positive and negative symptoms in schizophrenia | week11

SECONDARY OUTCOMES:
Specific Serum Immunological Parameters | baseline
  SGOT, SGPT, gamma-GT, BUN and creatinine
Specific Serum Immunological Parameters | week11
lipid profiles | based line, after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Band Lu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Ru-Band Lu, Tainan, Taiwan

REFERENCES:
- [Derived] Chen SL, Lee SY, Chang YH, Chen SH, Chu CH, Tzeng NS, Lee IH, Chen PS, Yeh TL, Huang SY, Yang YK, Lu RB, Hong JS. Inflammation in patients with schizophrenia: the therapeutic benefits of risperidone plus add-on dextromethorphan. J Neuroimmune Pharmacol. 2012 Sep;7(3):656-64. doi: 10.1007/s11481-012-9382-z. Epub 2012 Jun 23. PMID 22730040